CLINICAL TRIAL: NCT03817593
Title: The Assessment of Transcendental Meditation Training on ADD/ADHD Symptoms of Adolescents.
Brief Title: TM Meditation in Children With ADD/ADHD
Status: Withdrawn | Type: Observational
Why Stopped: Due to COVID epidemics and the multiple lock-downs, we were unable to begin the study
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Sheba-18-5309-DG-CTIL
Record Dates: First submitted 2019-01-07; First posted 2019-01-25 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Attention-Deficit Disorder in Adolescence
Keywords: meditation; heart rate variability; ADD; ADHD; children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Meditation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transcendental Meditation (TM): Each participant will have an individual instruction for 1 hour, followed by a course of 3 weekly group meetings (1-1.5 hours) The students shall meditate in a group for 10 minutes, twice a day, during 3 months, under the supervision of school teachers who will be instructed in TM technique.
  To ensure the quality of practice, a group follow-up will be performed 10 days after a completion of the course, and then each participant will receive personal meetings with TM instructor on a weekly basis during the first month, and twice a month for the second and third months.
  After additional 3 months participants in this group will be examined again, to assess sustainability of the effect
  Interventions: Other: Transcendental Meditation (TM)
- controls: Control group - Treatment as usual (TAU)

INTERVENTIONS:
Other: Transcendental Meditation (TM) — Each participant will have an individual instruction for 1 hour, followed by a course of 3 weekly group meetings (1-1.5 hours) The students shall meditate in a group for 10 minutes, twice a day, during 3 months, under the supervision of school teachers who will be instructed in TM technique.
  Groups: Transcendental Meditation (TM)

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common developmental disorders experienced in childhood, with limited options for effective pharmacological treatment. Transcendental Meditation (TM) has been proposed to be used as a tool for attentional training and modulating autonomic nervous system activity in the ADHD population. However, the empirical support in favor of meditation for ADHD is limited, and the mechanism by which TM may have an effect on ADD/ADHD is not understood. There is also a conflicted data as to the nature of autonomic dysregulation of ADHD.

Heart Rate Variability (HRV) represents the beat to beat changes of heart rate in the interbeat interval, and considered to be a non-invasive tool to study autonomic nervous system. There is evidence that a non-directive meditation may increase parasympathetic activity and overall HRV. To the best of our knowledge, the differential effect of meditation on ADHD symptoms: according to the baseline HRV of the participants, or ADHD subtypes has not been assessed.

The aim of this study is to collect the data on ADHD adolescents who will get TM training as a part of out-of-school program, which is offered all children diagnosed with ADD/ADHD, aged 11.5 y-16y, in the community center of Kadima-Zoran, Israel.

The assessment of all of the children participating in this program will be performed with the help of validated questionnaires for diagnosis and follow-up of ADD/ADHD, and HRV monitoring.

In order to perform an assessment in a controlled way, the instruction of TM shall take place in two cycles of 3 months each.

DETAILED DESCRIPTION:
Attention-deficit/hyperactivity disorder (ADHD) is one of the most common developmental disorders experienced in childhood, with a prevalence of 5 -10%, and can persist into adulthood (1) It is characterized by a combination of overactive, poorly modulated behavior with marked inattention and may involve physical aggression, which may be associated with a number of structural and functional abnormalities in the central nervous system (2).

Pharmacological treatment is often the treatment of choice; however its effectiveness is limited and often involves considerable side effects (3).

Meditation has been proposed to be used as a tool for attentional training and modulating autonomic nervous system activity in the ADHD population. A systematic review of meditation- based interventions for children with ADHD could not reach definite conclusions regarding their efficacy due to poor methodological quality of the studies (4).

A pilot randomized controlled study published few years ago demonstrated that three months of TM practice resulted in significant improvement of ADHD symptoms (5).

The mechanism by which TM may have an effect on ADD/ADHD is not understood. Furthermore, it is not clear whether TM may have a differential effect on the two subclasses of this condition: inattentive- and hyperactive- type

Individuals with ADHD probably have imbalances in autonomic nervous system activity, which may be associated with impairment of sustained attention (6) and emotional regulation (7,8,9).

Heart Rate Variability (HRV) represents the beat to beat changes of heart rate in the interbeat interval, resulting from dynamic balance of sympathetic and parasympathetic inputs to the heart being a non-invasive tool to study autonomic nervous system, has been proposed to be related to cognitive performance (10) and be a potential marker of stress (11). A lower resting HRV has been associated with greater difficulties in emotional regulation, especially a lack of emotional clarity and impulse control (12), depression and anxiety states (15), while higher levels - with higher cognitive performance, increased emotional regulation and perception of well-being (13, 14).

There is however no agreement as to the nature of autonomic dysregulation of ADHD (9,16,17).

The effect of meditation on autonomic nervous system via changes in heart rate variability has been studied recently. Interestingly, some of the techniques were associated with lower HRV (18), while others - with increased parasympathetic activity and HRV (19). To the best of our knowledge, the differential effect of meditation on ADHD symptoms: according to the baseline HRV of the participants, or ADHD subtypes has not been assessed.

Aims

Primary objective:

To collect the data on ADHD adolescents who will get TM training

Secondary objectives:

1. To assess whether improvement of symptoms may be sustained for 3 months after the intervention.
2. To assess whether the effect of TM on ADHD symptoms may be correlated with the baseline HRV or ADHD subtypes of the participants.

Participants and Methods

Study design TM classes are going to take place in the facility of Community Center at the Kadima Zoran Community Center for Culture and Sport (as an out-of-school program): a group of TM instructors will provide TM teaching to the adolescents with ADD/ADHD of the Zoran school, with the consent of the teachers and the parents of the children.

Since March 2019, the TM classes will be offered to all children aged 11.5 y-16y, with a confirmed diagnosis of ADD/ADHD, under supervision of the school teachers.

About 50 adolescents out of 60 adolescents, diagnosed with ADHD shall participate in this program.

The assessment and follow-up on these children will be performed by pediatric neurologist and HRV monitoring.

The instruction of TM shall be in two groups (of 20-30 children each). TM training for each group shall be 3 months. The children in both groups shall be followed up for 6 months, and assessed by the same parameters.

Participants:

About 50 adolescents out of 60 adolescents, diagnosed with ADHD who study at this school, are expected to participate in this program.

A senior pediatric neurologist will examine the children, confirm the diagnosis, according to the DSM 5 criteria, and shall obtain a written informed consent for the evaluation of the children during this program.

Current pharmacological treatment, ADHD subtype (e.g. inattentive type, combined type or mixed type) and the comorbidities will be documented.

Group 1

Two certified teachers of TM will teach these children according to the following protocol, as previously described by Grosswald et al(20):

Each participant will have an individual instruction for 1 hour, followed by a course of 3 weekly group meetings (1-1.5 hours) The students shall meditate in a group for 10 minutes, twice a day, during 3 months, under the supervision of school teachers who will be instructed in TM technique.

A group follow-up will be performed 10 days after a completion of the course, and then each participant will receive personal meetings with TM instructor on a weekly basis during the first month, and then twice a month.

After additional 3 months participants in this group will be examined again, to assess sustainability of the effect.

Group 2 Following the completion of the first 3 months period, the second group will receive TM training as above, and during the first 3 months this will be a reference (control) group.

Data analysis

The data will be analyzed according to the treatment groups. Similarly to the previous study (20) the expected statistical power of 93%will be calculated for comparison of means (Student T-test) .The assumed difference between groups is 0.1 and adopted Standard Deviation within the groups is ±0.1 (20).

Additional observations will be assessed according to the baseline HRV (sympathetic or parasympathetic predominance) and the ADHD subgroups (inattentive or hyperactive predominance), while the two ADHD subgroups and two HRV subgroups will be assessed independently with dichotomous outcomes. In the probable case that the two TM groups (A&B) shall not be significantly different, both groups may br assessed as one cohort with n=50, assuming dichotomous outcomes. This project may provide a preliminary assessment of the impact of ADHD subtype and of baseline HRV on the differential effect of TM on ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children with a confirmed diagnosis of ADHD

Exclusion Criteria:

* Comorbidities of Conduct Disorder, ODD, OCD
* Children on psychiatric medications
* Other chronic diseases

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: About 50 adolescents out of 60 adolescents, diagnosed with ADHD who study at at the Kadima Zoran School, Israel shall participate in this program.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Achenbach Youth Self-Report (YSR) assesses overall behavioral and emotional functioning. | The changes in scoring of this questionnaire from the baseline will be evaluated at the beginning of the study (time 0), after 3 months of TM instruction and after additional 3 months
  A self-reported scale that assesses overall behavioral and emotional functioning. appropriate behaviors, as well as inappropriate ones. The scale is designed for both parents and teachers, contains both social competency and behavior problem items.
Cardiac vagal tone - indexed by heart rate variability (HRV) | The changes in HRV from the baseline will be evaluated at the beginning of the study (time 0), after 3 months of TM instruction and after additional 3 months
  HRV refers to changes in normal cardiac interbeat intervals, are under control of the vagus nerve (21), may be a biomarker of psychopathology (22) and of faster recovery from stress (23). HRV is also linked to social and emotional function and can be seen as an objective measure of emotional and social functioning both in healthy and ill population (24).

SECONDARY OUTCOMES:
Conners 3 questionnaire | The changes in scoring of this questionnaire from the baseline will be evaluated at the beginning of the study (time 0), after 3 months of TM instruction and after additional 3 months
  Assesses cognitive, behavioral, and emotional problems, with a focus on ADHD and comordbid disorders-providing teacher, parent, and student perspectives
Behavior Rating Inventory of Executive Function (BRIEF) | The changes in scoring of this questionnaire from the baseline will be evaluated at the beginning of the study (time 0), after 3 months of TM instruction and after additional 3 months
  Assesses executive function behaviors in the school and home environments. The questionnaire was developed for parents and teachers of school-age children and is designed to assess the abilities of a broad range of children and adolescents. Tthe BRIEF is useful when working with children who have learning disabilities and attention disorders, traumatic brain injuries, lead exposure, pervasive developmental disorders, depression, and other developmental, neurological, psychiatric, and medical conditions.